CLINICAL TRIAL: NCT03905343
Title: Ribociclib-endocrine Combination Therapy Versus Chemotherapy as 1st Line Treatment in Patients With Visceral Metastatic Breast Cancer. A Multicenter, Randomized Phase III Trial.
Brief Title: Ribociclib-endocrine Combination Therapy Versus Chemotherapy as 1st Line in Visceral mBC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Feasibility (low patient accrual and financial reasons)
Sponsor: Swiss Cancer Institute (Other)
Collaborators: The Belgian Society of Medical Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 21/18; 2018-003648-22 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-04-05 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; Visceral metastatic breast cancer; Ribociclib; Ribociclib-endocrine
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Intervention Model Description: This is an international, multicenter, open-label, randomized phase III trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: endocrine therapy + ribociclib (Experimental)
  Interventions: Drug: Ribociclib; Other: Endocrine-Therapy
- B: mono-chemotherapy (Active Comparator)
  Interventions: Other: Mono-chemotherapy

INTERVENTIONS:
Drug: Ribociclib — Ribociclib 600mg p.o. d1-21, q4w in combination with endocrine treatment for 3 years.
  Arms: A: endocrine therapy + ribociclib
Other: Mono-chemotherapy — mono-chemotherapy for at least 12 weeks (afterwards, maintenance endocrine therapy ± ribociclib inhibitor is allowed) and up to 3 years.
  Arms: B: mono-chemotherapy
Other: Endocrine-Therapy — The choice of endocrine therapy is up to the investigator, but the chosen endocrine therapy has to be registered to be used in combination with ribociclib in the investigated indication.
  Arms: A: endocrine therapy + ribociclib

SUMMARY:
The aim of this trial is to assess if patients treated with the combination of ribociclib and endocrine therapy respond to treatment as fast as patients treated with chemotherapy only, without decreasing their quality of life (QoL).

DETAILED DESCRIPTION:
Breast cancer is the most frequent malignancy in women and the leading cause of cancer mortality in most countries in Europe. Metastatic breast cancer remains an incurable disease with a median overall survival (OS) of 2-4 years and a 5-year survival of only 25%. Patients with hormone receptor (HR)-positive breast cancer involving visceral disease at diagnosis have an even worse outcome.

Many oncologists still prefer to treat visceral disease primarily with chemotherapy rather than with endocrine treatment, thinking to receive a faster response with chemotherapy than with endocrine therapy, especially in patients with clinical symptoms or potentially threatening lesions. However, results from cross-sectional clinical practice studies suggest that endocrine therapy is associated with better quality of life, fewer concerns about side effects, less activity impairment and higher treatment satisfaction compared to chemotherapy. In addition, with the new data of CDK4/6 inhibitors combined with endocrine treatment there is an even better efficacy data available compared to endocrine therapy alone.

The aim of this trial is to assess if patients treated with the combination of ribociclib and endocrine therapy respond to treatment as fast as patients treated with chemotherapy only, without decreasing their quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to national law and ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically or cytologically confirmed diagnosis of HR-positive (ER+ ≥10%), HER2-negative advanced stage breast cancer
* Measurable visceral disease according to RECIST v1.1. Visceral disease in liver and/or lung. Peritoneal and/or pleural metastases only are accepted, with the condition to be measurable
* No previous systemic anticancer therapy for metastatic disease allowed
* Mono-chemotherapy is a reasonable treatment option
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before randomization and the patient has no evidence of disease at randomization. Less than 2 years is acceptable for adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* Patients with asymptomatic and stable (treated or untreated) central nervous system (CNS) metastases are eligible, provided they meet the following criteria:

  * ≤ 5 CNS lesions with a maximum diameter of the largest lesion of 10 mm
  * No evidence of progression at registration compared to the latest brain imaging (if applicable)
  * No ongoing requirement for corticosteroids as therapy for CNS disease
* Baseline QoL and pain questionnaires have been completed within 21 days prior to registration
* Postmenopausal women (without ovarian function suppression)
* Age ≥ 18 years
* WHO performance status 0-2
* Adequate bone marrow function: neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 90 g/L
* Adequate hepatic function: bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST ≤ 2.5 x ULN, AP ≤ 2.5 x ULN
* Adequate renal function: estimated glomerular filtration rate (eGFR) > 40 mL/min/1.73m2 (according to CKD-EPI or MDRD formula)
* Patient is able and willing to swallow trial drug as whole tablet

Exclusion Criteria:

* Visceral crisis (clinical judgment of treating investigator based on the ABC consensus: "visceral crisis is defined as severe organ dysfunction as assessed by signs and symptoms, laboratory studies, and rapid progression of disease. Visceral crisis is not the mere presence of visceral metastases, but implies important visceral compromise leading to a clinical indication for a more rapidly efficacious therapy, particularly since another treatment option at progression will probably not be possible")
* Symptomatic brain metastases indicative of active disease (defined as new and/or progressive brain metastases at the time of study entry) or leptomeningeal disease
* Any prior systemic anti-cancer treatment for advanced stage breast cancer
* Prior treatment with adjuvant CDK4/6 inhibitor
* Concurrent or recent (within 30 days of randomization) treatment with any other experimental drug. Exception: participation in SAKK 96/12 is allowed
* Concomitant use of other anti-cancer drugs or radiotherapy, except for local pain control
* Planned surgery of metastatic sites in the first 12 treatment weeks
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia)
* Electrocardiogram (ECG) abnormalities of Q-wave infarction (unless identified ≥ 6 months prior to randomization), or QTc interval >450 msec. The use of concomitant medications with a known significant risk of prolonging the QT interval or inducing Torsades de pointes is not allowed
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved national product information
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Quality of life-adjusted early disease control | at 12 weeks.
  A patient will be counted as a success for this endpoint when during the first 12 weeks
  - the response according to RECIST v1.1 is stable disease or better.
Quality of life-adjusted early disease control | at 12 weeks.
  A patient will be counted as a success for this endpoint when during the first 12 weeks
  - the QoL according Functional Assessment of Cancer Therapy-Breast Trial Outcome Index [FACT-B TOI] score does not worsen by 5 points or more.

SECONDARY OUTCOMES:
Disease Control (DC) at 12 weeks | week 6, 12.
  A patient will be counted as a success for this endpoint when during the first 12 weeks the response according to RECIST v1.1 is stable disease or better. Patients with missing response assessments within the first 12 weeks will be counted as failure unless there was no progressive disease (PD) documented within the first 12 weeks and the first subsequent assessment also shows no PD
Objective response rate (ORR) | week 6, 12, then every 12 weeks up to 3 years or end of trial treatment.
  ORR is defined as the proportion of patients having achieved complete response (CR) or partial response (PR) during trial treatment. Response will be evaluated according to RECIST v1.1 criteria.
Time to objective response (OR) | week 6, 12, then every 12 weeks up to 3 years or end of trial treatment.
  Time to OR will be calculated from randomization until first documented CR or PR according to RECIST v1.1 criteria. Time to OR will be calculated for patients having achieved a CR or PR at any time during trial treatment.
Progression-free survival (PFS) | week 6, 12, then every 12 weeks up to 3 years.
  PFS is defined as the time from randomization until progression according the RECIST v1.1 criteria or death from any cause, whichever occurs first. Patients not having an event at the time of analysis as well as patients starting a new anti-cancer therapy in the absence of an event will be censored at the date of their last tumor assessment before starting a new anti-cancer treatment, if any.
Time to treatment failure (TTF) | week 6, 12, then every 12 weeks up to 3 years.
  TTF is defined as the time from randomization until stopping of trial treatment from any cause. Patients not having an event at the time of analysis will be censored at the date of their last known date of trial treatment.
Overall survival (OS) at 3 years | week 6, 12, then every 12 weeks up to 3 years.
  OS at 3 years is determined by the Kaplan-Meier estimator for OS at 3 years. OS is defined as time from randomization to death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Changes in overall QoL (FACT-B) until 24 months | Changes from baseline to 24 months
  Changes in Functional Assessment of Cancer Therapy-Breast (FACT-B) total score (score range 0-148, higher scores indicate better quality of life)
Time to QoL deterioration | From baseline to 24 months
  Time to QoL deterioration is defined as the duration between baseline and first occurrence of a decrease of ≥ 5 points in the FACT-TOI score.
Time to QoL improvement | From baseline to 24 months
  Time to QoL improvement is defined as the duration between baseline and first occurrence of an increase of ≥ 5 points in the FACT-TOI score.
Time to pain improvement | From baseline to 24 months
  Improvements in pain will be assessed up to 24 months by the item pain severity of the Brief Pain Inventory (BPI), scale range: 0= no pain to 10 = pain as bad as one can imagine.
Adverse events (AEs) | every 4 weeks up to 3 years.
  All AEs will be assessed according to NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruhstaller, Prof, Study Chair — Kantonsspital St. Gallen - Breast Center St. Gallen
Locations (34):
- Austria (4):
  - Med. Univ. Klinik Graz, Graz
  - Tirol Kliniken - BrustGesundheitZentrum Tirol, Innsbruck
  - Salzburger Landeskliniken - Universitätsklinikum Salzburg, Salzburg
  - Universitätsklinik für Frauenheilkunde, Vienna
- Belgium (8):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Grand Hôpital de Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - CHC Mont Légia, Liège
  - CHU de Liege, Liège
  - CHR de la Citadelle, Liége
  - CHU UCL Namur - Site Sainte Elisabeth, Namur
  - Clinique-Saint-Pierre, Ottignies
- Switzerland (22):
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Brustzentrum Basel - Praxis für ambulante Tumortherapie, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Clinique des Grangettes, Chêne-Bougeries
  - Kantonsspital Graubuenden, Chur
  - Hôpital neuchâtelois, La Chaux-de-Fonds
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Lucerne
  - Hirslanden Klinik St. Anna Luzern, Lucerne
  - Onkologie Zentrum Spital Männedorf, Männedorf
  - Kantonsspital Olten, Olten
  - Brustzentrum Ostschweiz, Sankt Gallen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hôpital de Sion, Sion
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Brustzentrum, Winterthur
  - Onkologie Bellevue, Zurich
  - OnkoZentrum Zürich AG - Klinik im Park, Zurich
  - Universitäts Spital Zürich, Zurich